CLINICAL TRIAL: NCT04156802
Title: Project Relief: Developing Brain Stimulation as a Treatment for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00061967
Record Dates: First submitted 2019-11-04; First posted 2019-11-08 (Actual); Results first posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain; Chronic Lower Back Pain; Back Pain; Opioid Use; Opiate Dependence; Pain, Chronic; Neuropathic Pain; Chemotherapy-induced Peripheral Neuropathy
Keywords: Transcranial Magnetic Stimulation; Brain Stimulation; Treatment; Neuroimaging; Alternative
MeSH Terms: conditions — Chronic Pain; Back Pain; Opioid-Related Disorders; Neuralgia

STUDY DESIGN:
Intervention Model Description: This randomized, double-blind, sham-controlled study will parametrically evaluate the longitudinal effects of 16 days of rTMS to the MC (Aim 1) or the MPFC (Aim 2) on self-reported pain and the brain's response to pain. This will be done in a cohort of patients recruited from Wake Forest University clinics and the outer community with chronic lower back pain that may or may not be using prescription opiates for 3 or more months without adequate pain relief. Participants will be randomized to receive TMS to the MC, MPFC,or sham (50% at each site), using a Latin square randomization. Resting state connectivity will be collected. Quantitative Pain Testing will be collected 11 times. MRI data will be collected 3 times: before the 1st visit of TMS, after the 12th visit of TMS, and after the 16th visit of TMS.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Real TBS to the mPFC (Experimental): Two sessions of real Theta Burst Stimulation (TBS) will be delivered to the medial prefrontal cortex (mPFC) over the course of the treatment and maintenance phase of the study
  Interventions: Device: Real TBS to the mPFC
- Sham TBS to the mPFC (Sham Comparator): Two sessions of sham Theta Burst Stimulation (TBS) will be delivered to the medial prefrontal cortex (mPFC) over the course of the treatment and maintenance phase of the study
  Interventions: Device: Sham TBS to the mPFC
- Real TBS to the MC (Experimental): Two sessions of real Theta Burst Stimulation (TBS) will be delivered to the somatomotor cortex (MC) over the course of the treatment and maintenance phase of the study
  Interventions: Device: Real TBS to the MC
- Sham TBS to the MC (Sham Comparator): Two sessions of sham Theta Burst Stimulation (TBS) will be delivered to the somatomotor cortex (MC) over the course of the treatment and maintenance phase of the study
  Interventions: Device: Sham TBS to the MC

INTERVENTIONS:
Device: Real TBS to the mPFC — This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded)
  Arms: Real TBS to the mPFC
Device: Sham TBS to the mPFC — This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded). The MagVenture MagPro system has an integrated active sham that passes current through two surface electrodes placed on the skin beneath the coil.
  Arms: Sham TBS to the mPFC
Device: Real TBS to the MC — This will be delivered with the Magventure Magpro system (double blinded).
  Arms: Real TBS to the MC
Device: Sham TBS to the MC — This will be delivered with the Magventure Magpro system (double blinded). The MagVenture MagPro system has an integrated active sham that passes current through two surface electrodes placed on the skin beneath the coil.
  Arms: Sham TBS to the MC

SUMMARY:
Effective control of chronic pain is a top priority in the United States, as approximately 10% of adults have severe chronic pain most of which is chronic lower back pain (CLBP). However, despite the advances in neuroscience over the past 20 years, chronic pain is largely treated with opiate narcotics, much as was done in the Civil War. In addition to their high abuse liability and dependence potential, only 30 40% of chronic pain patients declare they receive satisfactory (>50%) relief from their pain through pharmacological treatment. In these patients a common clinical practice is to escalate the dose of opiates as tolerance develops which unfortunately has contributed to escalation in opiate overdose deaths, a resurgence of intravenous heroin use, and $55 billion in societal costs. Consequently, there is a critical need for new treatments that can treat pain and reduce reliance on opiates in individuals with chronic pain.

The proposed study will be the first to employ a randomized, double-blind, sham-controlled design to parametrically evaluate the longitudinal effects of 16 days of Repetitive transcranial magnetic stimulation (rTMS) to the primary motor cortex (MC) or the medial prefrontal cortex (MPFC) on self-reported pain and the brain s response to pain. This will be done in a cohort of patients recruited from the community as well as Wake Forest Baptist Health (WFBH) clinics with chronic lower back pain that have not been able to find adequate pain relief, whether or not they are using prescription opiates for 3 or more months. Participants will be randomized to receive rTMS to the MC, MPFC, or sham (50% at each site), using a Latin square randomization. Resting state connectivity will be collected 3 times: before the 1st day of TMS, after the 12th day of TMS, and before the 16th day of TMS (the last day administered).

DETAILED DESCRIPTION:
Effective control of chronic pain is a top priority in the United States, as approximately 10% of adults have severe chronic pain - most of which is chronic lower back pain (CLBP). However, despite the advances in neuroscience over the past 20 years, chronic pain is largely treated with opiate narcotics, much as was done in the Civil War. In addition to their high abuse liability and dependence potential, only 30-40% of chronic pain patients declare they receive satisfactory (>50%) relief from their pain through pharmacological treatment. In these patients a common clinical practice is to escalate the dose of opiates as tolerance develops - which unfortunately has contributed to escalation in opiate overdose deaths, a resurgence of intravenous heroin use, and $55 billion in societal costs. Consequently there is a critical need for new, treatments that can treat pain and reduce reliance on opiates in individuals with chronic pain.

The goal of this proposal is to evaluate 2 novel non-invasive brain stimulation strategies to mitigate pain and the brain's response to pain in CLBP patients that are currently taking chronic opiates, or that are seeking an alternative treatment for pain. Transcranial Magnetic Stimulation (TMS), can induce long term potentiation (LTP-like) and long term depression (LTD-like) effects on brain activity in a frequency dependent manner. Our group has previously demonstrated that LTP-like TMS to the dorsolateral prefrontal cortex (DLPFC, a node in the Executive Control Network (ECN)) can decrease perceived pain and corresponding blood oxygen level dependent (BOLD) signal in the "Pain Network'. The Pain Network is an expansion of the Salience Network (SN; insula, dorsal anterior cingulate) which includes the thalamus and somatosensory cortex. The analgesic effects of DLPFC TMS can be blocked by naloxone - suggesting that the analgesic effects of LTP-like DLPFC TMS are opiate mediated. Additionally, DLPFC TMS delivered postoperatively leads to less patient administered morphine use (PCA-pump) in the hospital and less opiate use in the outpatient setting. These data all suggest that LTP-like DLPFC TMS is a promising candidate for treating pain.

An alternative strategy is to apply LTD-like stimulation to the medial prefrontal cortex (LTD-like mPFC rTMS. This strategy is based on our understanding of functional neural architecture, wherein the SN is modulated by 2 other core networks: the executive control network (ECN) and the default mode network (DMN). As stated above, it is possible to attenuate activity in the SN through LTP-like TMS to the DLPFC, a node in the ECN. It is also possible to attenuate the SN through LTD-like TMS to the ventral medial prefrontal cortex (a node in the DMN). The proposed study will be the first to employ a randomized, double-blind, sham-controlled design to parametrically evaluate the longitudinal effects of 16 days of rTMS to the MC or the MPFC on self-reported pain and the brain's response to pain. This will be done in a cohort of patients recruited from the community as well as WFBH clinics with chronic lower back pain that have not been able to find adequate pain relief, whether or not they are using prescription opiates for 3 or more months. Participants will be randomized to receive rTMS to the MC, MPFC, or sham (50% at each site), using a Latin square randomization. Resting state connectivity will be collected 3 times: before the 1st day of TMS, after the 12th day of TMS, and before the 16th day of TMS (the last day administered).

Aim 1. Evaluate MC rTMS as a tool to dampen pain and the engagement of the Pain Network. Hypothesis 1: MC TMS will attenuate the baseline brain response to pain (Pain Network activity) and increase activity in the ECN when the patient is given instructions to 'control' the pain.

Aim 2. Evaluate MPFC rTMS as a tool to dampen pain and the engagement of the Pain Network. Hypothesis 1: MPFC TMS will also attenuate the baseline brain response to pain (Pain Network activity) but will not effect the ECN or SN when the patient is given instructions to 'control' the pain.

(Exploratory Aim): The investigator will evaluate if there are rate-dependent effects between baseline SN connectivity with the ECN and DMN and the efficacy of each TMS strategy on subjective pain. Data will be analyzed by using multivariate pattern analysis (MVPA). While the primary outcomes will be magnetic resonance imaging (MRI) Visit 1 versus Visit 2, the investigator will also examine the relative 'durability' of the effects on pain by comparing the MRI data at the end of all TMS visits between and within groups with factor analysis.

The relative efficacy of these strategies will directly translate to development of a large clinical trial investigating rTMS as an innovative, new treatment option for pain in patients with CLBP.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (to maximize participation)
2. Can currently be using prescription opiates
3. Able to read and understand questionnaires and informed consent.
4. Is not at elevated risk of seizure (i.e., does not have a history of seizures, is not currently prescribed medications known to lower seizure threshold)
5. Does not have metal objects in the head/neck.
6. Does not have a history of traumatic brain injury, including a head injury that resulted in hospitalization, loss of consciousness for more than 10 minutes, or having ever been informed that they have an epidural, subdural, or subarachnoid hemorrhage.
7. Does not have a history of claustrophobia leading to significant clinical anxiety symptoms.

Exclusion Criteria:

1. Any psychoactive illicit substance use (except marijuana and nicotine) within the last 30 days by self-report and urine drug screen.
2. Meets DSM V criteria for current axis I disorders of obsessive-compulsive disorder, bipolar affective disorder, schizophrenia, dissociate disorders, eating disorders, and any other psychotic disorder or organic mental disorder.
3. Has current suicidal ideation or homicidal ideation.
4. Has the need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications and medications for ADHD.
5. Females of childbearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.
6. Has current charges pending for a violent crime (not including DUI related offenses).
7. Does not have a stable living situation.
8. Suffers from chronic migraines.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merideth A Addicott, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. All data is de-identified.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Real TBS to the mPFC | Sham TBS to the mPFC | Real TBS to the MC | Sham TBS to the MC
Started | 13 | 6 | 13 | 6
Completed | 9 | 5 | 10 | 5
Not Completed | 4 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real TBS to the mPFC | Sham TBS to the mPFC | Real TBS to the MC | Sham TBS to the MC | Total
Number analyzed (Participants) | 13 | 6 | 13 | 6 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (13) | 62 (9) | 63 (7) | 59 (8) | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 6 | 4 | 22
  Male | 4 | 3 | 7 | 2 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 5 | 1 | 8
  White | 11 | 6 | 8 | 5 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Patient Reported Pain and Discomfort
Description: The investigators expect changes in self reported qualitative pain assessment via a numeric pain rating scale when comparing active vs sham. Pain rating values will be assessed and reported through the duration of the study. Percent change from baseline values ranged from -100 to 500. Larger, positive values represent increased pain and worse outcomes.
Time Frame: From Baseline to the last follow up session (16 weeks)
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Real TBS to the mPFC | Sham TBS to the mPFC | Real TBS to the MC | Sham TBS to the MC
Number analyzed (Participants) | 9 | 5 | 10 | 5
percent change from baseline | 47 (190) | 13 (32) | -30 (39) | -18 (28)

2. Other Pre Specified Outcome: Changes in Pain Thresholds Using the Quantitative Pain Testing (QST) Task, Which Utilizes Pressure From the Medoc Pathway Algomed Device to Detect Pain Thresholds
Description: Based on pilot data, the investigators expect an interaction between treatment (Real DLPFC or MPFC TMS vs. Sham) and time (Before vs. After rTMS) on reported painfulness using a quantitative sensory testing technique determines the sensation and pain thresholds of warm temperatures. Painfulness ratings will be assessed and reported through the duration of the study.
Time Frame: Through study completion, an average of 4 and a half months
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Neuroimaging Outcomes: Changes in the Brain's Response to Pain as Specified by Changes in BOLD Signal
Description: Evaluating real and sham iTBS to the motor cortex vs. real and sham iTBS to the medial prefrontal cortex and how the brain activity attenuates the baseline brain response to pain (Pain Network activity). It is predicted that regardless of which site, TBS in general will dampen pain and the engagement of the Pain Network when compared to baseline activity before any treatment (as measured through BOLD signal).
Time Frame: Through study completion, an average of 4 and a half months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment until final follow-up session, 16 weeks.
Arm/Group | Real TBS to the mPFC | Sham TBS to the mPFC | Real TBS to the MC | Sham TBS to the MC
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6 | 0/13 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/6 | 0/13 | 0/6
Other Adverse Events (participants affected / at risk) | 5/13 | 1/6 | 2/13 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real TBS to the mPFC (N=13) | Sham TBS to the mPFC (N=6) | Real TBS to the MC (N=13) | Sham TBS to the MC (N=6)
Headache (General disorders) | 5 (14) | 1 (2) | 2 (4) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT04156802/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT04156802/ICF_000.pdf